CLINICAL TRIAL: NCT04731610
Title: Randomized, Multicenter, Phase III Trial to Assess Conformal Post-operative Radiotherapy vs. Surveillance After Complete Resection of Stage II/III Thymoma
Brief Title: Randomized, Multicenter, Phase III Trial to Assess Conformal Post-operative Radiotherapy vs. Surveillance After Complete Resection of Stage II/III Thymoma (RADIO-RYTHMIC-01)
Acronym: RADIO-RYTHMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2020-09
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Thymoma Malignant Recurrent
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-operative radiotherapy (Other): Tumour resection followed by radiotherapy.
  Interventions: Other: Radiotherapy
- Surveillance after tumour resection (Other): Tumour resection
  Interventions: Other: Surveillance after resection

INTERVENTIONS:
Other: Radiotherapy — postoperative radiotherapy after complete resection of thymoma
  Arms: Post-operative radiotherapy
Other: Surveillance after resection — Surveillance after tumour resection
  Arms: Surveillance after tumour resection

SUMMARY:
The primary objective of the study : to compare the Recurrence-Free survival (RFS) between arms. RFS is defined as time from randomisation to the first recurrence (either local-regional or distant) or death of any cause.

ELIGIBILITY:
Inclusion Criteria:

1. 18 < Age < 75 years old
2. ECOG performance status ≤1
3. Preoperative chemotherapy is allowed. Maximum of 4 cycles are authorized. Surgery should be realized ≤ 2 months after the last chemotherapy injection.
4. Histologically diagnosed thymoma at pathological examination of surgical specimen after pathological review; for note, centralized, real-time, systematic pathological review is standard through the RYTHMIC network in France
5. Complete resection at pathological examination of the surgical specimen after surgery conducted through standard, recommended approach ensuring accurate assessment of resection status
6. Stage IIb or III disease according to the Masaoka-Koga staging system; this corresponds to stage pT1a with capsule invasion, until stage pT3 N0 M0 in the 8th TNM staging system TNM UICC/AJCC
7. Availability of thoracic Computed-Tomography (CT) scan with IV contrast (in the absence of contra-indications) or PET scan performed before surgery
8. Availability of a thoracic Computed-Tomography (CT) scan with IV contrast (in the absence of contra-indications) showing absence of residual disease after surgical resection of the tumor
9. Pulmonary function tests after surgery with FEV1 ≥ 1L or ≥ 35% of the theoretical value and DLCO ≥ 40%
10. Signature of informed consent form

Exclusion Criteria:

- 1. Age > 75 years old 2. Histology of thymic carcinoma 3. Delivery of post-operative chemotherapy, concurrent chemotherapy to radiotherapy 4. Presence of microscopic or macroscopic residual tumor after surgery or metastases (R1 or R2 resection) 5. Uncontrolled, clinically significant pleural or pericardial effusion 6. Patients with prior radiation therapy to the thorax. Patients treated with conformal radiotherapy for prior breast or head and neck neoplasms should be discussed with PI 7. Evidence of severe or uncontrolled systemic disease as judged by the investigator 8. Recent (< 6 months) severe cardiac disease (uncontrolled arrhythmia, congestive heart failure, infarction, pace-maker) or pulmonary disease. Controlled and non clinically symptomatic arrhythmia is allowed.

9. Current or past history of neoplasm diagnosed within the last 3 years, except: basal cell carcinoma of the skin, in situ carcinoma of the cervix, and bladder in situ. A patient diagnosed for another neoplasm 3 years ago or more, treated and considered as cured may be included in the study if all the other criteria are respected 10. Pregnancy or breast feeding or inadequate contraceptive measures for women of childbearing potential during PORT 11. Patients who, for family, social, geographic or psychological reasons, cannot be adequately followed up and/or are incapable of undergoing regular controls, 12. Patients deprived of freedom or under guardianship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2031-12-28 (Estimated); Study Completion 2032-12-28 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free survival (RFS) | 3 years
  to compare the Recurrence-Free survival (RFS) between arms. RFS is defined as time from randomisation to the first recurrence (either local-regional or distant) or death of any cause.

SECONDARY OUTCOMES:
Local-regional (pleural or pericardial) recurrence | 3 years
  Local-regional (pleural or pericardial) recurrence; location of recurrence /removed

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU Caen, Caen
  - CLCC François BACLESSE, Caen
  - CLCC Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHU Lyon, Lyon
  - AP-HM Hôpital Nord, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat AP-HP, Paris
  - CHU Haut Lévêque, Pessac
  - CHU Rennes Hôpital Sud, Rennes
  - CHU Rouen, Rouen
  - CLCC Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CHU Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHRU Tours, Tours
  - Institut de Cancérologie de Lorraine Nancy, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets . Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).